CLINICAL TRIAL: NCT03973970
Title: Assessing the Ability of the T-SPOT®.TB Test to Identify Those at Risk of Active Mycobacterium Tuberculosis Infection Using the Normalized Tuberculosis (TB) Specific Lymphocyte Response.
Brief Title: Assessing the Ability of the T-SPOT®.TB Test (IQ)
Acronym: IQ
Status: Completed | Type: Observational
Sponsor: Oxford Immunotec (Industry)
Responsible Party: Sponsor
Other Study IDs: US TX 153
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-07

CONDITIONS: Tuberculosis
Keywords: TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells (PBMCs) and plasma will be retained and stored at the Lung Infection and Immunity laboratory Biobank for 3 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Arm 1- T-SPOT.TB assay: Test Arm 1: T-SPOT.TB test using density gradient isolation (Leucosep) For each subject recruited in the study, cells will be isolated using Leucosep Tubes and T-Cell Xtend reagent according to package insert. For each subject recruited in the study, the T-SPOT.TB assay will be run according to the assay package insert.
- Test Arm 2-QuantiFERON-TB Gold Plus assay: Test Arm 2: QuantiFERON-TB Gold Plus For each subject recruited in the study, the QuantiFERON-TB Gold Plus (QFT-Plus) assay will be run according to the assay package insert.

SUMMARY:
The primary objective of this clinical research study is to demonstrate performance of the normalized TB specific lymphocyte response (NTBSLR) in identifying patients with active TB disease. The secondary exploratory objective is to demonstrate that active TB cannot be identified using an antigen-to-mitogen ratio derived from an ELISA-based IGRA.

DETAILED DESCRIPTION:
This study will enroll up to 202 subjects (assumes 15 % exclusion/drop-out rate). The target number of subjects is 75 active TB (recruited from subjects presenting at TB clinics) and 100 active TB excluded (recruited from subjects in the community).

All subjects enrolled in this study will be men or women, aged 18 years or older.

Duration: 1 year

ELIGIBILITY:
Subject Inclusion Criteria: Cohort 1A and 1B

* Must be at least 18 years of age
* Must be able to provide informed consent
* Must be able to provide a minimum of 10 mL of whole blood at each visit
* Must be T-SPOT.TB positive
* First visit suspect TB subjects with no prior history of TB diagnosis Subject exclusion criteria: Cohort 1A and 1B
* Negative in the T-SPOT.TB test
* Previous or pre-existing confirmed TB diagnosis
* On anti-TB treatment for less than 1 week*
* Not meeting inclusion criteria

Subject inclusion criteria: Cohort 2A and 2B

* Must be at least 18 years of age
* Must be able to provide informed consent
* Must be able to provide a minimum of 10 mL of whole blood at each visit
* Must be T-SPOT.TB positive
* No prior history of TB diagnosis

Subject exclusion criteria: Cohort 2A and 2B

* Negative T-SPOT.TB test
* Previous or pre-existing confirmed TB diagnosis
* On anti-TB treatment
* Symptoms of active TB
* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and Female 18 years of age and older
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
NTBSLR | 2 year
  The primary objective of this study is to demonstrate performance of the normalized Tuberculosis (TB) specific lymphocyte response (NTBSLR) in identifying patients with active Tuberculosis (TB) disease.

SECONDARY OUTCOMES:
IGRA | 2 year
  The secondary exploratory objective is to demonstrate that active Tuberculosis (TB) cannot be identified using an antigen-to-mitogen ratio derived from an ELISA-based Interferon-Gamma Release Assay (IGRA).

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Restrepo, MD, Principal Investigator — UTHealth Houston, School of Public Health
Locations (1):
- University of Texas Health, Brownsville, Texas, United States

IPD SHARING:
Plan to Share IPD: No